CLINICAL TRIAL: NCT00201396
Title: A Multicenter Phase III Trial Comparing Induction Chemotherapy Followed by Concurrent Chemoradiotherapy Versus Concurrent Chemoradiotherapy Alone in Stage IV Nasopharyngeal Carcinoma (NPC)
Brief Title: A Multicenter Trial Comparing Induction C/T Followed by CCRT v.s. CCRT Alone in Stage IV Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Tri-Service General Hospital (Other); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); Chung Shan Medical University (Other); Changhua Christian Hospital (Other); Chi Mei Medical Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1303
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2006-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: A Multicenter Phase III Trial; Induction Chemotherapy; Concurrent Chemoradiotherapy; Stage IV Nasopharyngeal Carcinoma (NPC); randomization; disease-free survival
MeSH Terms: conditions — Nasopharyngeal Carcinoma

ARMS (2):
- A arm (Active Comparator): CCRT
  Interventions: Radiation: CCRT
- B arm (Experimental): Induction/CCRT
  Interventions: Radiation: CCRT; Drug: Mitomycin C,Epirubicin,Cisplatin,5-Fluorouracil,Leucovorin

INTERVENTIONS:
Radiation: CCRT — Radiation with weekly Cisplatin
Drug: Mitomycin C,Epirubicin,Cisplatin,5-Fluorouracil,Leucovorin — Induction C/T + CCRT
  Arms: B arm

SUMMARY:
Investigate the effect of induction MEPFL chemotherapy followed by concurrent chemoradiotherapy (CCRT) on the disease control and survival in treatment of patients with advanced NPC.

DETAILED DESCRIPTION:
Rationale of induction chemotherapy:

Distant metastasis is the major cause of treatment failure and deaths in patients with loco-regionally advanced NPC.

Concurrent chemoradiotherapy may prolong survivals for patients with advanced NPC, but it is still flawed by high incidence of distant metastasis.

Induction chemotherapy with MEPFL has been shown to reduce the incidence of distant metastasis in a Phase II study.

Induction chemotherapy plus concurrent chemoradiotherapy may improve the survival of patients with advanced NPC.

Objectives:

Investigate the effect of induction MEPFL chemotherapy followed by concurrent chemoradiotherapy (CCRT) on the disease control and survival in treatment of patients with advanced NPC.

Study design:

This is a randomized, multi-center Phase III study. Patients will be randomized to CCRT with or without the MEPFL induction chemotherapy.

Type and number of patients:

Patients with stage IVA (T4) and/or IVB (N3) but without distant metastasis will be enrolled. A total of up to 480 patients will be randomized to detect an improvement of median overall survival from 5.8 to 8.7 years, with an a=0.05 and power of 0.8 using a two-sided logrank test with one interim analysis.

Treatment schedule:

Induction chemotherapy and CCRT:

Arm A: Weekly cisplatin concurrently with radiotherapy Arm B: Induction MEPFL three cycles followed with weekly cisplatin concurrently with radiotherapy.

Study endpoints:

The primary endpoint is the disease-free survival that will be calculated as the duration between the date of randomization and the date of recurrence of NPC at any site including persistent disease after +induction chemotherapy/CCRT, or death from any cause (failed), or the date of withdrawal (last contact date, censored), or the scheduled data analysis date (censored).( revised 8/27/2004)

ELIGIBILITY:
Inclusion Criteria:

* Histologically proved nasopharyngeal carcinoma.
* T4NxM0 or TxN3M0 disease by UICC/AJCC 1997 staging system. (30)
* Eastern Cooperative Oncology Group performance status < 2.
* A leukocyte count ≥3750/mL, Hb ≥ 10 g/dL, and a platelet count ≥100,000/mL.
* A serum bilirubin level < 1.5 mg/dL, serum creatinine level < 1.6 mg/dL or creatinine clearance > 60 mL/min.
* Age less than 70 years old
* An informed consent signed.

Exclusion Criteria:

* Evidence of metastatic disease.
* Presence of another malignancy other than treated squamous/basal cell carcinoma of the skin.
* Presence of uncontrolled hypertension, poorly controlled heart failure.
* Presence of active infection.
* Patients who have been or are being treated with chemotherapy, radiotherapy, immunotherapy, or other experimental therapies.
* Women who test positive for pregnancy.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2003-08; Primary Completion 2009-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the disease-free survival. | 10 years
  follow up for 2 years after off study treatment

SECONDARY OUTCOMES:
Secondary endpoints include overall survival and tumor response rate. | 10 years
  follow up for 2 years after off study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Long Hong, MD, PhD, Principal Investigator — Taiwan cooperative oncology group
Locations (4):
- Taiwan (4):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang-Gung Memorial Hospital(Lin-Kou),, Taoyuan District

REFERENCES:
- [Derived] Hong RL, Hsiao CF, Ting LL, Ko JY, Wang CW, Chang JTC, Lou PJ, Wang HM, Tsai MH, Lai SC, Liu TW. Final results of a randomized phase III trial of induction chemotherapy followed by concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in patients with stage IVA and IVB nasopharyngeal carcinoma-Taiwan Cooperative Oncology Group (TCOG) 1303 Study. Ann Oncol. 2018 Sep 1;29(9):1972-1979. doi: 10.1093/annonc/mdy249. PMID 30016391
- See also: Related Info — http://english.nhri.org.tw/inst_cancer/ca_TCOGresearch.php